CLINICAL TRIAL: NCT06139796
Title: Pharmacokinetics, Safety and Acceptability of a Solid Paediatric Fixed-dose Combination of Darunavir/Ritonavir (DRV/r) 120/20 mg for Children Living With HIV
Brief Title: Pharmacokinetics Safety and Acceptability of DRV/r for Children Living With HIV
Acronym: UNIVERSAL2
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study not started as the IMP is re-worked by the manufacturer
Sponsor: PENTA Foundation (Network)
Collaborators: AMS-PHPT Research Collaboration (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Mère et Enfant de la Fondation Chantal Biya (Other); Centre Hospitalier National d'Enfants Albert Royer (Unknown); University of Zimbabwe Clinical Research Centre (UZCRC) (Unknown); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIVERSAL2
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections
Keywords: HIV; Darunavir; Ritonavir; Paediatrics; new formulation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Open-label, multi-centre, single-arm, phase I/II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A Twice daily (Experimental): DRV/r twice daily (BID): 30 children with 1 or 2 DRV RAM* weighing 10 to <25 kg (10 per weight band: 10-13.9kg, 14-19.9kg, 20-24.9kg)
  Interventions: Drug: DRV/r FDC (120/20mg)
- Cohort B Once daily (Experimental): DRV/r once daily (OD): 20 children with no DRV RAM* weighing 10 to <20 kg (10 per weight band: 10-13.9kg, 14-19.9kg)
  *DRV RAMs: V11I, V32I, L33F, I47V, I50V, I54M, I54L, T74P, L76V, I84V and L89V
  Interventions: Drug: DRV/r FDC (120/20mg)

INTERVENTIONS:
Drug: DRV/r FDC (120/20mg) — Initiation of DRV/r FDC (120/20mg) as part of antiretroviral therapy (ART) with an Optimized Background Therapy (OBT)

SUMMARY:
The UNIVERSAL2 study is a research project designed to evaluate a newly developed formulation of an approved drug for children living with HIV aged over 3 years and weighing between 10 and 25 kg. The aim of UNIVERSAL2 is to determine the right dosage of this new formulation.

DETAILED DESCRIPTION:
The UNIVERSAL2 study is a research project designed to evaluate a newly developed formulation of an approved drug for children living with HIV aged over 3 years and weighing between 10 and 25 kg. The aim of UNIVERSAL2 is to determine the right dosage of this new formulation.

It is a combination of two anti-HIV medicines called darunavir (DRV) and ritonavir (RTV). The DRV/RTV combination is well known and has been used for a long time in adults and children to treat HIV infection but there is no combined pediatric formulation that has been adapted to the needs of children ("child friendly" formulation).

The new combination has been developed in the form of fixed-dose combination tablets with a dose of 120 mg of DRV and 20 mg of RTV (DRV/RTV 120/20) in each tablet. Depending on their weight and the need to take the medication once or twice a day, children may receive 2, 3 or 4 DRV/RTV 120/20 tablets at any given time.

The aim of UNIVERSAL2 is to determine the correct dosage and to assess the safety and acceptability of the new drug for children living with HIV.

The study will focus on two groups of children.

* Group A will include children with one or two specific viral genetic mutations linked to DRV resistance and will receive DRV/RTV twice daily.
* Group B will include children without DRV resistance viral gene mutations who will receive DRV/RTV once daily.

All children will start taking the DRV/r at the beginning of the study. After two weeks, participants will be invited to stay at the clinic for blood samples to be taken at different times of the day in order to understand how the drug is absorbed, metabolised and excreted in the body (pharmacokinetic tests). They will then continue to be monitored at the clinic several times over a 24-week period, with additional blood tests to be sure children are tolerating the drug well and that it helps to control HIV replication. Participants and their carers will also be asked to answer some questions to determine how acceptable the new tablets are to children and carers.

ELIGIBILITY:
Inclusion Criteria:

* • Confirmed HIV-1 infection

  * Aged ≥ 3 years
  * With unsuppressed viral load (HIV-1 RNA viral load > 1000 c/mL) on ART-regimen and eligible to switch to new DRV/r 120/20 mg-based regimen per investigator's judgement
  * Able to swallow the 120/20 mg DRV/r tablets
  * Willing to receive the 120/20 mg DRV/r tablets
  * Parents or guardians, and children where appropriate, willing and able to give informed consent and to adhere to the protocol
  * Cohort-specific inclusion criteria:

Cohort A:

* Have 1 or 2 DRV resistance-associated mutations (RAMs)*
* Weigh 10 to <25 kg at screening

Cohort B:

* Have no DRV RAMs*
* Weigh 10 to <20 kg at screening. *DRV RAMs: V11I, V32I, L33F, I47V, I50V, I54M, I54L, T74P, L76V, I84V and L89V

Exclusion Criteria:

* Presence of >2 darunavir RAMs*

  * Failure of protease genotypic resistance testing at baseline, except if treatment history indicates that it is very unlikely
  * Resistance to all NRTI available in the country or impossibility to define an OBT
  * Intercurrent illness (enrolment can take place after the illness resolves)
  * Creatinine ≥ 1.8 Upper Limit of Normal (ULN) or ALT ≥ 5 ULN or (ALT ≥ 3 ULN and bilirubin ≥2 ULN) at screening.
  * Severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices, or persistent jaundice), or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
  * History or presence of known allergy or other contraindication to DRV/r or their components as described in the Summary of Product Characteristics (SmPC)
  * Concomitant medications that may interact with the current antiretroviral treatment, in particular TB drugs (i.e: rifampicin, rifabutin, rifapentine, …).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Darunavir | From enrollment to the end of treatment at 24 weeks
  area under the concentration-time curve (AUC0-12) (Cohort A)
Pharmacokinetics Darunavir | From enrollment to the end of treatment at 24 weeks
  area under the concentration-time curve (AUC0-24) (Cohort B)
Pharmacokinetics Darunavir | From enrollment to the end of treatment at 24 weeks
  maximum plasma concentration (Cmax)
Pharmacokinetics Darunavir | From enrollment to the end of treatment at 24 weeks
  12 hours or 24 hours post dose concentrations (C12 or C24)
Safety events | From enrollment to the end of treatment at 24 weeks
  serious adverse events (SAEs)
Safety events | From enrollment to the end of treatment at 24 weeks
  adverse events (AEs) of Grade 3 or higher
Safety events | From enrollment to the end of treatment at 24 weeks
  treatment related AEs
Safety events | From enrollment to the end of treatment at 24 weeks
  AEs leading to treatment discontinuation or modification

SECONDARY OUTCOMES:
Acceptability | From enrollment to the end of treatment at 24 weeks
  Questionnaire
Efficacy of treatment | From enrollment to the end of treatment at 24 weeks
  HIV-1 RNA <50 c/mL and <400 c/mL
Efficacy of treatment | From enrollment to the end of treatment at 24 weeks
  Occurrence of a new or recurrent WHO clinical stage 3 or 4 event
Efficacy of treatment | From enrollment to the end of treatment at 24 weeks
  Change in CD4 cell count and percentage from baseline to week 24
Pharmacokinetics Ritonavir | From enrollment to the end of treatment at 24 weeks
  RTV PK parameters and DRV unbound concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Albert Faye, Study Chair — Hôpital Robert Debré and Université Paris Cité
Locations (5):
- Centre Mère et Enfant de la Fondation Chantal Biya, Yaoundé, Cameroon, Cameroon
- Centre Hospitalier National d'Enfants Albert Royer, Dakar, Senegal, Senegal
- Uganda (2):
  - Baylor College of Medicine Children's Foundation, Kampala, Uganda
  - Joint Clinical Research Centre (JCRC), Kampala
- University of Zimbabwe Clinical Research Centre (UZCRC), Harare, Zimbabwe, Zimbabwe

IPD SHARING:
Plan to Share IPD: No